CLINICAL TRIAL: NCT06489054
Title: Effects of a Peer-based Educational Project on Adolescents' Oral Health Literacy
Brief Title: Effects of Peer-based Education on Adolescent Oral Health Literacy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Paulo Frazao, Professor (Full), University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FSP-USP
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Health Literacy
Keywords: Health Education, Dental; Adolescent
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Experimental group and control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer education (Experimental): An initial assessment will be carried out to determine the socioeconomic, demographic profile and dental data and baseline data on literacy and attitudes related to oral health through questionnaires, after which participants will be invited to participate in a cycle of oral health education activities for three months on the experimental group (peer-based education). After the experimental stage, the literacy and attitudes questionnaires related to oral health will be reapplied, so that a comparative analysis can be carried out within and between groups.
  Interventions: Other: Peer education
- Conventional education (Active Comparator): An initial assessment will be carried out to determine the socioeconomic, demographic profile and dental data and baseline data on literacy and attitudes related to oral health through questionnaires, after which participants will be invited to participate in a cycle of oral health education activities for three months on the control group (dentist lecture). After the experimental stage, the literacy and attitudes questionnaires related to oral health will be reapplied, so that a comparative analysis can be carried out within and between groups.
  Interventions: Other: Conventional education

INTERVENTIONS:
Other: Peer education — An initial assessment will be carried out to determine the socioeconomic, demographic profile and dental data and baseline data on literacy and attitudes related to oral health through questionnaires, after which participants will be invited to participate in a cycle of oral health education activities for three months on the experimental group (peer-based education). After the experimental stage, the literacy and attitudes questionnaires related to oral health will be reapplied, so that a comparative analysis can be carried out within and between groups.
  Arms: Peer education
Other: Conventional education — An initial assessment will be carried out to determine the socioeconomic, demographic profile and dental data and baseline data on literacy and attitudes related to oral health through questionnaires, after which participants will be invited to participate in a cycle of oral health education activities for three months on the control group (dentist lecture). After the experimental stage, the literacy and attitudes questionnaires related to oral health will be reapplied, so that a comparative analysis can be carried out within and between groups.
  Arms: Conventional education

SUMMARY:
This project aims to identify whether an oral health peer education strategy can influence the level of functional literacy and oral health attitudes of adolescents aged 15 to 19 years. An experimental study will be carried out, a non-randomized controlled community trial, with two groups of educational strategy in oral health: peer education (experimental group) and conventional education (control group). For data collection, three questionnaires will be applied: for socioeconomic, demographic and dental data; assessment of oral health literacy (BOHL-AQ); and assessment of oral health attitudes; the last two being applied before and after the intervention.

DETAILED DESCRIPTION:
This project aims to identify whether an oral health peer education strategy can influence the level of functional literacy and oral health attitudes of adolescents aged 15 to 19 years. An experimental study will be carried out, a non-randomized controlled community trial, carried out in the municipality of Araruna-PB, with two groups of educational strategy in oral health: peer education (experimental group) and conventional education (control group). For data collection, three questionnaires will be applied: for socioeconomic, demographic and dental data; assessment of oral health literacy (BOHL-AQ); and assessment of oral health attitudes; the last two being applied before and after the intervention. Descriptive analysis will be performed and a test will be applied to assess the normality of the data. The psychometric properties of the BOHL-AQ with adolescents will be evaluated using factor analysis. For literacy and attitude data, a comparison of means before and after the intervention will be performed using the intragroup paired and unpaired Student t test. All analyzes will be performed using the Statistical Package for the Social Sciences (SPSS) 25.0, considering a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 15 to 19 years old, who obtain consent from their parents/guardians (for those under 18 years of age), voluntarily accept to participate in the study and are present on the day the questionnaires are administered.

Exclusion Criteria:

* Adolescents with physical and/or mental disabilities that make it impossible to follow the activities proposed in the intervention and respond to the questionnaires.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Oral health literacy | The first data collection (baseline) occurred 2 months after participant recruitment and the second collection will be after the intervention, 3 months after baseline.
  A specific questionnaire, Brazilian Oral Health Literacy-Adults Questionnaire - BOHL-AQ, will be used to measure oral health literacy before and after the oral health education intervention.

SECONDARY OUTCOMES:
Attitudes related to oral health | The first data collection (baseline) occurred 2 months after participant recruitment and the second collection will be after the intervention, 3 months after baseline.
  A questionnaire will be used to measure attitudes related to oral health before and after the oral health education intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Frazão, Study Director — University of Sao Paulo; Helene Moura, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No